CLINICAL TRIAL: NCT00892788
Title: A Behavioral Intervention for Reducing Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: UCHC/Storrs and Regional Campus Incentive Grants (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-128-1; 20090200 (Other Grant/Funding Number: UCHC/Storrs and Regional Campus Incentive Grants)
Record Dates: First submitted 2009-04-03; First posted 2009-05-05 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Contingency Management
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Participants assigned to Group A will receive the LEARN (Lifestyle, Exercise, Attitudes, Relationships, Nutrition) Program weight loss manual and will be instructed to read a section of the manual each week and complete suggested activities. They will also meet with the research staff once a week for weigh-in and supportive counseling.
  Interventions: Behavioral: weight loss manual-guided individual therapy sessions
- B (Experimental): Participants assigned to Group B will receive the LEARN manual and will meet with research staff each week for weigh-in and supportive counseling. They will also receive contingency management or the opportunity to earn draws with the chance of winning prizes for losing weight and completing healthy activities.
  Interventions: Behavioral: contingency management; Behavioral: weight loss manual-guided individual therapy sessions

INTERVENTIONS:
Behavioral: contingency management — Prize-based contingency management for weight loss
  Arms: B
Behavioral: weight loss manual-guided individual therapy sessions — once weekly counseling sessions with research staff

SUMMARY:
This study will examine a contingency management (CM) intervention designed to provide incentives for losing weight versus participating in a manual-guided behavioral weight loss intervention alone. Participants in the CM condition will earn the opportunity to win prizes by losing weight and completing activities that contribute to weight loss, such as keeping daily food and physical activity diaries, choosing healthy foods, exercising, and using other weight loss strategies. The investigators will determine if the CM improves weight loss relative to the usual care manual-guided intervention alone.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* body mass index in kg/m2 (BMI) between 30.0 and 39.9
* seated blood pressure of 100/60-140/90 mmHg
* ability to speak English and read at the 6th grade level
* willingness to be randomly assigned to one of two groups

Exclusion Criteria:

* any serious acute or chronic medical problems that may impact dietary or exercise regimens or impact weight loss
* psychiatric exclusions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
absolute and relative weight loss | Weeks 1-12
changes in waist circumference | Week 1 and Week 12
proportion of participants achieving clinically significant weight loss (5% or more of baseline weight) | Week 1 and Week 12

SECONDARY OUTCOMES:
indices of treatment retention | Weeks 1-12
changes on measures of diet quality, physical activity, and physiological parameters such as blood pressure, lipoproteins, insulin, and glucose levels | Week 1 and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States